CLINICAL TRIAL: NCT07326995
Title: A Phase 2 Clinical Study to Evaluate the Safety and Efficacy of PA9159 Inhalation Aerosol for the Treatment of Adult Bronchial Asthma
Brief Title: Safety and Efficacy of PA9159 Inhalation Aerosol for the Treatment of Adult Bronchial Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Palo Alto Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA9159AS-201
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PA9159 60 μg (Experimental): Fifteen subjects will be randomly assigned to receive 60 μg of PA9159 Metered-Dose Inhaler for 28 days. Subjects will be administered three vials of drug (Inhaler bottle A ,Inhaler bottle B and Inhaler bottle C) Twice a day: In the morning, take 2 puffs from Bottle A and 2 puffs from Bottle B. In the evening, take 4 puffs from Bottle C.
  Interventions: Drug: PA9159 Metered-Dose Inhaler, 60 μg per day for 28 days
- PA9159 120 μg (Experimental): Fifteen subjects will be randomly assigned to receive 120 μg of PA9159 Metered-Dose Inhaler for 28 days. Subjects will be administered three vials of drug (Inhaler bottle A ,Inhaler bottle B and Inhaler bottle C) Twice a day: In the morning, take 2 puffs from Bottle A and 2 puffs from Bottle B. In the evening, take 4 puffs from Bottle C.
  Interventions: Drug: PA9159 Metered-Dose Inhaler, 120 μg per day for 28 days
- PA9159 240 μg (Experimental): Fifteen subjects will be randomly assigned to receive 240 μg of PA9159 Metered-Dose Inhaler for 28 days. Subjects will be administered three vials of drug (Inhaler bottle A ,Inhaler bottle B and Inhaler bottle C) Twice a day: In the morning, take 2 puffs from Bottle A and 2 puffs from Bottle B. In the evening, take 4 puffs from Bottle C.
  Interventions: Drug: PA9159 Metered-Dose Inhaler, 240 μg per day for 28 days
- placebo (Placebo Comparator): Fifteen subjects will be randomly assigned to receive placebo Metered-Dose Inhaler for 28 days. Subjects will be administered three vials of drug (Inhaler bottle A ,Inhaler bottle B and Inhaler bottle C) Twice a day: In the morning, take 2 puffs from Bottle A and 2 puffs from Bottle B. In the evening, take 4 puffs from Bottle C.
  Interventions: Drug: Placebo Metered-Dose Inhaler without PA9159, Twice daily for 28 days

INTERVENTIONS:
Drug: PA9159 Metered-Dose Inhaler, 60 μg per day for 28 days — PA9159 of 60 μg is delivered orally through a metered-dose Inhaler , Twice daily for 28 days.
  Arms: PA9159 60 μg
Drug: PA9159 Metered-Dose Inhaler, 120 μg per day for 28 days — PA9159 of 120 μg is delivered orally through a metered-dose Inhaler , Twice daily for 28 days.
  Arms: PA9159 120 μg
Drug: PA9159 Metered-Dose Inhaler, 240 μg per day for 28 days — PA9159 of 240 μg is delivered orally through a metered-dose Inhaler , Twice daily for 28 days.
  Arms: PA9159 240 μg
Drug: Placebo Metered-Dose Inhaler without PA9159, Twice daily for 28 days — Placebo is delivered orally through a metered-dose Inhaler , Twice daily for 28 days.
  Arms: placebo

SUMMARY:
PA9159 is a highly potent novel corticosteroid. The purpose of this study is to evaluate the safety, efficacy and characteristics of population pharmacokinetics of multiple dosing of PA9159 Inhalation Aerosol in patients with bronchial asthma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel, placebo-controlled clinical trial. Subjects of 60 with bronchial asthma are planned to be included in this study. With a ratio of 1: 1: 1: 1 to be randomized allocated to receive PA9159 Inhaler of 60 μg, 120 μg, and 240 μg, or placebo, with 15 subjects in each group. The duration of this study is approximately 42 days, including screening, baseline, treatment observation, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years inclusive, regardless of gender;
* According to the definition in the Chinese "Guidelines for Prevention and Treatment of Bronchial Asthma (2020 Edition)," subjects diagnosed with bronchial asthma, including those with an initial diagnosis of asthma, or those diagnosed with asthma during childhood or adolescence with stable condition who have not received long-term treatment but exhibit significantly more pronounced symptoms in adulthood and/or recently compared to the past;
* Pre-randomization, pulmonary function tests show 60% ≤ FEV1% predicted ≤ 85%;
* Any objective test result indicating variable airflow limitation conducted within 1 year prior to screening is positive, or the bronchodilator test during the screening period is positive, i.e., an increase in FEV1 ≥ 12% and an absolute increase in FEV1 ≥ 200 mL 15-30 minutes after inhaling 400 μg salbutamol (if the bronchodilator test result does not meet the positive threshold, a repeat bronchodilator test is allowed within 14 days after the test [excluding the test day]); or the bronchial provocation test is positive, i.e., a decrease in FEV1 ≥ 20% after inhaling a provocant (methacholine or histamine); or the average daily diurnal variability of peak expiratory flow (PEF) (calculated as the sum of daily PEF diurnal variability over 7 consecutive days divided by 7) > 10%;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Subjects who are unable to correctly use a nebulizer, cannot tolerate nebulized inhalation administration, or fail inhalation administration training;
* Subjects with other pulmonary diseases, including chronic obstructive pulmonary disease, bronchiectasis, pulmonary fibrosis, tuberculosis, etc., for which, in the investigator's judgment, asthma remains the dominant condition;
* Coexistence of other clinically significant conditions that may affect lung function, including but not limited to pleural diseases, mediastinal diseases, diaphragmatic disorders, myasthenia, thoracic deformities, etc.;
* History of severe cardiovascular diseases, such as congestive heart failure, coronary artery disease, myocardial infarction, arrhythmia, uncontrolled hypertension (resting seated systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg on two or more consecutive measurements), etc., which, in the investigator's judgment, would put the subject at risk or may affect the interpretation of study results;
* Subjects with hyperthyroidism, assessed by the investigator as unsuitable for participation in this trial;
* History of severe hematologic, hepatic, psychiatric, renal, or other diseases that, in the investigator's judgment, would put the subject at risk or may affect the interpretation of study results;
* History of malignancy within the past five years (excluding cured cervical intraepithelial neoplasia, thyroid cancer, or basal cell carcinoma of the skin diagnosed and cured within 5 years);
* Subjects who have undergone or are expected to undergo solid organ or bone marrow transplantation within the next year;
* Hypokalemia (serum potassium < 3.5 mmol/L during screening);
* Type I diabetes or poorly controlled Type II diabetes (fasting blood glucose > 11.1 mmol/L during screening);
* Known or pre-randomization examination revealing oral, pharyngeal, or esophageal candidiasis;
* Abnormal liver or kidney function during screening (ALT and/or AST > 2× upper limit of normal; Scr > 1.5× upper limit of normal);
* Positive hepatitis B surface antigen or hepatitis B core antibody with HBV DNA ≥ 2000 IU/mL, positive hepatitis C antibody with HCV RNA ≥ 1000 IU/mL, positive human immunodeficiency virus antibody, or history of acquired immunodeficiency syndrome;
* Known allergy to any component of inhaled corticosteroids or salbutamol preparations;
* Respiratory tract infection, sinus infection, or acute otitis media within 4 weeks before screening or during the run-in period, which, in the investigator's judgment, would lead to changes in asthma treatment or affect the subject's asthma status;
* Asthma exacerbation requiring systemic corticosteroid treatment within 4 weeks before screening or during the run-in period, or asthma requiring oral corticosteroid therapy, or other conditions requiring systemic corticosteroid treatment;
* Use of strong CYP3A4 enzyme inhibitors (e.g., ritonavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, saquinavir, ketoconazole, telithromycin, etc.) within 4 weeks before dosing, or need for concomitant use of strong CYP3A4 inhibitors during the trial;
* Smoking cessation < 1 year at screening (including cigarettes, cigars, pipe tobacco, e-cigarettes, etc.), or previous smoking history > 10 pack-years [pack-years = number of packs per day × years of smoking, where 1 pack = 20 cigarettes];
* History of drug abuse, substance abuse, or alcoholism within 2 years before screening [alcoholism defined as average daily alcohol intake > 2 units (1 unit = 360 mL beer, or 45 mL of 40% alcohol liquor, or 150 mL wine)];
* Pregnant or lactating women, or women planning pregnancy during the trial;
* Subjects who have participated in other clinical trials within 1 month before screening;
* Any other reason considered by the investigator to make the subject unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation the change in morning pre-dose forced expiratory volume in one second (FEV1) from baseline to week 4 of treatment. | From pre-dose until 28 days post-dose
  After the subject takes a deep breath as much as possible, the volume of air that can be exhaled in the first second when exhaling with maximum force and speed. This is one of the most core indicators in pulmonary function tests, directly reflecting the patency of the airways (especially the large airways). A lower FEV₁ value indicates more severe airway obstruction. Therefore, the difference is calculated as the value after 28 days of treatment minus the baseline value. A larger upward change indicates more significant symptom improvement.

SECONDARY OUTCOMES:
Evaluation the change from baseline in pre-dose FEV1 at week 1 and week 2 of treatment. | From pre-dose until 14 days post-dose
Evaluation the change from baseline in pre-dose morning and evening peak expiratory flow (PEF) at weeks 1, 2, and 4 of treatment. | From pre-dose until 28 days post-dose
Proportion of patients with asthma exacerbations during the treatment period. | From pre-dose until 28 days post-dose
Proportion and frequency of patients using rescue medication over the 4-week treatment period. | From pre-dose until 28 days post-dose
Evaluation the change from baseline in the Asthma Control Test (ACT) score after 4 weeks of treatment. | From pre-dose until 28 days post-dose
Evaluation the change from baseline in the Asthma Quality of Life Questionnaire (AQLQ) score at weeks 2 and 4 of treatment. | From pre-dose until 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zuo, Principal Investigator — The First Affiliated Hospital of Nanchang University
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No